CLINICAL TRIAL: NCT05929261
Title: Stress Response to Virtual Exposure to Risky Movements After Anterior Cruciate Ligament (ACL) Rehabilitation and Its Relationship With Kinesiophobia
Brief Title: Stress Response to Virtual Risky Movement Exposure and Kinesiophobia After Anterior Cruciate Ligament (ACL) Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ogun Koyagasioglu, MD, PhD Candidate, Director of the project, Ege University
Other Study IDs: 22-12.2Tl31
Record Dates: First submitted 2023-06-15; First posted 2023-07-03 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Kinesiophobia; Anterior Cruciate Ligament Injuries
Keywords: Kinesiophobia; Anterior Cruciate Ligament Injuries; Virtual Reality; Stress; Athlete; Sports Medicine
MeSH Terms: conditions — Kinesiophobia; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Study group will be examined for outcome measurements.
- Control Group: Control group will be examined for outcome measurements.

SUMMARY:
In this study, patients who have completed their rehabilitation after Anterior Cruciate Ligament (ACL) reconstruction surgery will be examined with physiological stress response test while being exposed to risky athletic movements via virtual reality headsets. In the next, step patients' functional performance tests will be examined and their relation with stress responses will be examined.

ELIGIBILITY:
Inclusion Criteria for Study Group:

* 18 years or older
* Male gender
* Having history of isolated unilateral ACL reconstruction surgery
* Physician clearance for unrestricted physical activity after having at least 6-months of rehabilitation following surgery
* Willing to return to sports that require cutting and landing motions
* Not having any sports injuries past three months
* Not having any previous orthopaedic surgery other than ACL reconstruction surgery

Inclusion Criteria for Control Group:

* 18 years or older
* Male gender
* Playing sports that require cutting and landing motions
* Physician clearance for unrestricted physical activity
* Not having any sports injuries past three months
* Not having any previous orthopaedic surgery

Exclusion Criteria for Study Group:

* Having a reinjury during rehabilitation
* Having multiple ligament injuries before the surgery
* Diagnosed with knee osteoarthritis
* Diagnosed with knee cartilage injury
* Diagnosed with meniscus tear

Exclusion Criteria for Control Group:

* Diagnosed with ACL injury
* Diagnosed with knee osteoarthritis
* Diagnosed with knee cartilage injury
* Diagnosed with meniscus tear

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study group consists of subjects who had ACL reconstruction surgery and willing to return to sports activities.
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Subjective Kinesiophobia Status - Anterior Cruciate Ligament - Return to Sport after Injury (ACL-RSI) scale | From 0 to 6 months
  ACL-RSI scale evaluates psychological readiness to return to sports participation after ACL reconstruction and has items related to fear of reinjury/accidental injury during sport activities.
  The scale contains 12 questions and each question is scored from 0 to 100 in 10-point increments according to the visual analog scale. The scale score is calculated by adding the scores from all 12 questions and dividing by 12. A high score on the scale indicates a positive psychological response.
Physiological Stress Responses - Heart Rate Variability (HRV) Metrics | From 0 to 6 months
  Metrics will be measured with Shimmer 3 GSR Development and Consensys GSR Development Kit. Low Frequency (LF), High Frequency (HF), Low Frequency to High Frequency ratio (LF/HF), root mean square of successive differences (RMMSD) will be measured from participants while watching stress evoking videos. Metrics will be measured according to the Task Force guidelines in 1996. RMSSD reflects the integrity of vagus nerve-mediated autonomic control of the heart, HF reflects parasympathetic activity, and LF is proportional to sympathetic activity but influenced by parasympathetic tone. LF/HF reflects sympathetic activity dominancy over parasympathetic activity.
Physiological Stress Responses - Galvanic Skin Response (GSR) Metrics | From 0 to 6 months
  Metrics will be measured with Shimmer 3 GSR Development and Consensys GSR Development Kit. Skin conductance response (SCR) will be measured from participants while watching stress evoking videos. SCR is the measurement of the electrical conductivity of the skin and represents the activation of sweat glands in response to a particular stressor stimuli.
Functional Tests Landing Error Scoring System (LESS) score | From 0 to 6 months
  Participants will be tested for their landing with a standardized jump-landing from a box task. Subjects will jump down from the box and land on the ground and then immediately jump vertically upward as high as possible. We will rate for every participant by observing in both the sagittal and the frontal plane of jump- landing technique while the subject was in contact with the ground after landing from the box.
  Scoring will be made as "No" (0 points) and "Yes" (1 point) for Items 1-15. For Item16, it will be evaluated as "Excellent" (0 points), "Average" (1 point) and "Hard" (2 points). For item 17, "Excellent" (0 points), "Average" (1 point) and "Bad" (2 points). The total score of 17 items will be evaluated. The higher the score obtained from the test result, the worse the jump landing. LESS scores will be interpreted in four different categories: excellent (LESS score <4), good (4<LESS score ≤5), moderate (5<LESS score ≤6), and poor (LESS score >6).
Functional Tests - Hop tests (single legged) | From 0 to 6 months
  Participants will be tested for leg hop tests which described in the literature by Ross et al. 2002. >10% difference between tested legs will be considered as asymmetry.
  Single Hop for Distance. Subjects will be instructed to hop as far as possible forward and land on the same leg. The distance from the starting line to the point where the subject is landed will be measured.
  Triple Hop for Distance. Subjects will be instructed to take 3 maximal hops forward with the designated leg. The distance from the starting line to the point where the subject is landed will be measured.
  Crossover Hop for Distance. Subjects will be instructed to take 3 maximal hops while crossing over a line each time. The distance from the starting line to the point where the subject is landed will be measured.
  Six Meter Hop for Time. Subjects will be instructed to hop 6m distance as quickly as possible with the designated leg. Time will be measured from start to the time the subject crossed the finish line.
Functional Tests - T-test | From 0 to 6 months
  For each participant, a running t test will be performed, which will evaluate their agility during running with changes of direction. Participants will be asked to run forward for 10 m, then change to side-steps to the right for 5 m, then 10 m of side-steps to the left, followed by 5 m of side- steps to the right, ending with 10 m of backwards running. Three repetitions will be performed at maximum speed and the average time for the three repetitions will be calculated.
  Completing the test in less than 11 seconds will be classified as high agility, and finishing in 11 seconds or more will be classified as low agility.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No